CLINICAL TRIAL: NCT00913315
Title: Efficacy Study of Tamsulosin and Tolterodine Treatment of Men With Chronic Prostatitis/Chronic Pelvic Pain Syndrome and Lower Urinary Tract Symptoms
Brief Title: Efficacy Study of Tamsulosin and Tolterodine Treatment for Chronic Prostatitis
Acronym: ESTTFCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Collaborators: Fuling Central Hospital of Chongqing City (Other)
Responsible Party: Yong Chen, Urology department , Fuling Central Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQU023
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Prostatitis
Keywords: prostatitis; Adrenergic alpha-Antagonists; tolterodine
MeSH Terms: conditions — Prostatitis | interventions — Tolterodine Tartrate; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tolterodine + tamsulosin (Experimental)
  Interventions: Drug: tolterodine; Drug: tamsulosin
- tamsulosin + placebo (Active Comparator)
  Interventions: Drug: tamsulosin; Drug: placebo

INTERVENTIONS:
Drug: tolterodine — 4 mg of tolterodine ER
  Arms: tolterodine + tamsulosin
Drug: tamsulosin — 0.4 mg of tamsulosin once a day for 8 weeks
Drug: placebo — placebo once a day for 8 weeks
  Arms: tamsulosin + placebo

SUMMARY:
The purpose of this study is to determine whether tamsulosin and tolterodine are effective in the treatment of men with lower urinary tract symptoms and chronic prostatitis/chronic pelvic pain syndrome.

DETAILED DESCRIPTION:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is a common disorder in urological clinics. Most of the clinically CP/CPPS are to some extent associated with storage (irritative) symptoms, such as increased frequency, urgency, and nocturia, namely many patients with CP/CPPS have overactive bladder symptoms. Alpha-blocker therapy has been advocated as a treatment modality for CP/CPPS. Some trials showed a statistically and likely clinically significant treatment effect, while other trials showed no benefit. Therefore, tamsulosin combination with tolterodine treatment for CP/CPPS may be more effective than tamsulosin single.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of CP/CPPS based on the classification of US National Institutes of Health, aged 18-45 years
2. total score of at least 12 on the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI)
3. urinary score of at least 4 on the CPSI
4. subjects who anticipate improving symptoms

Exclusion Criteria:

1. previous treatment with any other alpha-adrenergic receptor blocker and antimuscarinic agents for symptoms of CP/CPPS or for any other reason
2. those who had had previous urinary tract infection with the last year
3. those who had been treat or were taking medication that could affect lower urinary tract function
4. those who met the criteria for chronic bacterial prostatitis after lower urinary tract localization studies
5. those who had other significant medical problems

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Chronic Prostatitis Symptom Index | 4 months

SECONDARY OUTCOMES:
Peak urinary flow rate | 4 months
International Index of Erectile Function | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chen, M.D., Principal Investigator — Chongqing Medical University
Locations (1):
- Department of Urology, the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Nickel JC, Krieger JN, McNaughton-Collins M, Anderson RU, Pontari M, Shoskes DA, Litwin MS, Alexander RB, White PC, Berger R, Nadler R, O'Leary M, Liong ML, Zeitlin S, Chuai S, Landis JR, Kusek JW, Nyberg LM, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network. Alfuzosin and symptoms of chronic prostatitis-chronic pelvic pain syndrome. N Engl J Med. 2008 Dec 18;359(25):2663-73. doi: 10.1056/NEJMoa0803240. PMID 19092152